CLINICAL TRIAL: NCT07086612
Title: Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) and Transverse Orthodontic Deficiency in Children
Acronym: ASCOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 761-ASCOT; 2025-A00478-41 (Other: ID RCB)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea; Transverse Maxillary Deficiency
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transverse deficiency maxilla (Experimental): patient with transverse deficiency maxilla
  Interventions: Diagnostic Test: over nigtht ventilatory polysomnograph test
- other type of maxilla deficiency (Other): patient with other type maxilla deficiency
  Interventions: Diagnostic Test: over nigtht ventilatory polysomnograph test

INTERVENTIONS:
Diagnostic Test: over nigtht ventilatory polysomnograph test — Every patient will have an overnight polysomnography test.

SUMMARY:
OSAHS (Obstructive Sleep Apnea Hypopnea Syndrome) in children is a frequent respiratory disorder, whose prevalence is estimated at between 1.2 and 5.7%, and which, if left untreated, can cause severe medical complications. This prevalence tends to be underestimated. Diagnosis is made following a clinical examination noting the presence of characteristic clinical and polysomnographic criteria. Multidisciplinary management has been widely described in the literature, and various therapeutic options have been indicated. Rapid maxillary expansion has proved highly effective in the treatment of this condition. This syndrome is a real public health problem and must be diagnosed as early as possible. Through our research, we would like to study whether there is a causal link between an orthodontic problem of the transverse direction and the presence of SAHOS in children. In other words, we would like to assess whether children who clinically present an orthodontic deficiency of their transverse dimension are more likely to develop SAHOS than children without this deficit. If this proves to be true, then a new clinical sign could enable certain healthcare professionals to detect this syndrome early, and be able to refer patients to physicians as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 6 and 16 years
* Patients with a transverse orthodontic deficiency (group "CAS")
* Patients with another type of orthodontic deficiency (group "CONTROL") such as tooth rotation, crowding, mild Angle Class II or Class III dental occlusion
* Patient who has given free, informed oral consent
* Patient whose legal representatives have given their free written consent
* Patient affiliated with a health insurance scheme

Exclusion Criteria:

* Patients refusing to participate in the study
* Patients whose legal representatives refuse to participate in the study

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
study whether children with a transverse orthodontic deficiency have a higher risk of developing Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) compared to those without this deficiency, | 1 months after enrollement
  compare the proportion of children with an Apnea-Hypopnea Index (AHI) >1, , based on the presence or absence of a transverse deficiency." AHI is evaluated with the polysomnography exam

SECONDARY OUTCOMES:
study whether all children with a transverse orthodontic deficiency systematically have Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) | one month after enrollement
  distribution of Apnea-Hypopnea Index (AHI) values among these children
Investigate a link between the severity of this transverse deficiency and the severity of OSAHS. | 1month after enrollement
  Distribution of AHI values among children based on the extent of the transverse deficiency. Three groups will be formed for the transverse deficiency : one for pure endognathies, one for endoalveolies, and one for crossbite occlusions.".
  AHI is evaluated with the polysomnography exam.
impact of hteSeverity of transferse deficiency on the snoring events frequency. | 1months after enrollement
  Average number of snoring events per hour based on the severity of the transverse deficiency. Three groups for the transverse defficiency will be formed: one for pure endognathies, one for endoalveolies, and one for crossbite occlusions.
  Number of snoring event will be mesured by the polysomnography exam.
diagnostic value of the sleep disorder screening scale for children aged 4 to 16 years | 1month after enrollement
  comparison of the sleep disorder screening scale results with the results of the polysomnography exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'orthopédie dento-cranio-maxillo faciale, Rouen, France

IPD SHARING:
Plan to Share IPD: No